CLINICAL TRIAL: NCT00707265
Title: A Prospective, Randomized Clinical Investigation of rhBMP-2 and Compression Resistant Matrix With the CD HORIZON® Spinal System for Posterolateral Lumbar Fusion in Patients With Symptomatic Degenerative Disc Disease
Brief Title: rhBMP-2/CRM/CD HORIZON® Spinal System Pivotal Study
Acronym: CRM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01-05
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Transplantation, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational (Experimental): Open bilateral posterolateral implantation of the rhBMP-2/CRM/CD HORIZON® Spinal System.
  Interventions: Device: rhBMP-2/CRM/CD HORIZON® Spinal System
- Control (Active Comparator): The bilateral posterolateral implantation of the autogenous bone harvested from the iliac crest with the CD HORIZON® Spinal System.
  Interventions: Device: Autograft/CD HORIZON® Spinal System

INTERVENTIONS:
Device: rhBMP-2/CRM/CD HORIZON® Spinal System — The rhBMP-2/CRM component of the investigational device consists of recombinant human Bone Morphogenetic Protein-2 (rhBMP-2) and a compression resistant matrix (CRM) carrier consisting of an absorbable collagen sponge imbedded with biphasic calcium phosphate.
  The posterior spinal fixation system, the CD HORIZON® Spinal System, is a commercially available rod-based spinal system intended for temporary stabilization of the spine in order to facilitate fusion. The CD HORIZON® Spinal System is available in either titanium or stainless steel. For this study, only titanium implant components will be used.
  Other Names: rhBMP-2; CRM; CD HORIZON® Spinal System
  Arms: Investigational
Device: Autograft/CD HORIZON® Spinal System — The control will be autogenous bone taken from the iliac crest of the patient and placed bilaterally across two adjacent transverse processes and used in conjunction with the CD HORIZON® Spinal System. When used as a posterior spine thoracic/lumbar system, the CD HORIZON® CANNULATED M8 MULTI-AXIAL SCREW components are intended for several indications including degenerative disc disease.
  Other Names: Autograft; CD HORIZON® Spinal System
  Arms: Control

SUMMARY:
The purpose of this study was to evaluate the rhBMP-2/CRM/CD HORIZON® Spinal System as a method of facilitating spinal fusion in patients with degenerative disc disease.

DETAILED DESCRIPTION:
This clinical trial was conducted to evaluate the rhBMP-2/CRM/CD HORIZON® Spinal System for posterolateral fusion treatment of patients with symptomatic degenerative disc disease versus the control group of autogenous bone with the CD HORIZON® Spinal System.

The investigational treatment was the open bilateral posterolateral implantation of the rhBMP-2/CRM/CD HORIZON® Spinal System. One investigational implant was placed across two adjacent transverse processes on each side of the spine during the spinal fusion procedure.

The control treatment was the bilateral posterolateral implantation of the autogenous bone harvested from the iliac crest with the CD HORIZON® Spinal System.

ELIGIBILITY:
Inclusion Criteria:

Each patient participating in this clinical trial must meet all of the following inclusion criteria:

1. Has degenerative disc disease as noted by back pain of discogenic origin, with or without leg pain, with degeneration of the disc confirmed by patient history of pain and radiographic studies:
2. Requires fusion of a single level disc space from L1 to S1.
3. Has not responded to non-operative treatment (e.g., bed rest, physical therapy, medications, spinal injections, manipulation, and/or TENS) for a period of 6 months.
4. If of child-bearing potential, patient is non-pregnant, non-nursing, and agrees to use adequate contraception for 1 year following surgery.

Exclusion Criteria:

A patient meeting any of the following criteria is to be excluded from this clinical trial:

1. Has primary diagnosis of a spinal disorder other than degenerative disc disease with Grade 1 or less spondylolisthesis at the involved level.
2. Had previous spinal fusion surgical procedure at the involved level.
3. Requires spinal fusion at more than one lumbar level.
4. Has been previously diagnosed with osteopenia.
5. Has presence of active malignancy or prior history of malignancy (except for basal cell carcinoma of the skin).
6. Has a history of autoimmune disease (e.g. Systemic Lupus Erythematosus or dermatomyositis).
7. Has a history of exposure to injectable collagen or silicone implants.
8. Has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP 2/CRM implantation.
9. Has received any previous exposure to any/all BMP's of either human or animal extraction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2002-03; Primary Completion 2005-05 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Overall Success | 24 months
  A patient will be considered an overall success if all of the following conditions are met:
  1. fusion;
  2. pain/disability (Oswestry) improvement;
  3. maintenance or improvement in neurological status;
  4. no serious adverse event classified as implant associated or implant/surgical procedure associated;
  5. no additional surgical procedure classified as a "failure."

SECONDARY OUTCOMES:
Fusion | 24 months
  Fusion is defined as:
  1. Evidence of bridging trabecular bone.
  2. No evidence of motion.
  3. Absence of cracking, as evidenced by radiolucent lines completely through the fusion mass.
Pain/Disability Status | 24 months
  The self-administered Oswestry Low Back Pain Disability Questionnaire will be used. Success will be defined as pain/disability improvement postoperatively according to the definition: Preoperative Score - Postoperative Score >= 15 points
Overall Neurological Status | 24 months
  Neurological status will be assessed preoperatively and postoperatively using a neurological status scale. Neurological status is based on four types of measurements (sections): motor, sensory, reflexes, and straight leg raise. Overall measure of neurological status will be based on success statuses in the four parameters.
General Health Status | 24 months
  The Medical Outcomes Study 36-item Short Form Health Survey (SF-36) will be used to assess general health status. The SF-36 results can be summarized into two components, a physical component summary (PCS) and a mental component summary (MCS). Success will be defined as a maintenance or improvement in status postoperatively as compared to the preoperative condition. To be classified as a success, the following criteria must be met:
  PCSPostop - PCSPreop >= 0; MCSPostop - MCSPreop >= 0
Back Pain | 24 months
  Numerical rating scales will be used to evaluate pain intensity and duration. The pain score (0 min, 20 Max) is derived by adding the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and duration scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Success for back and leg pain is described as follows:
  Preoperative Score - Postoperative Score >=0
Leg Pain | 24 months
  Numerical rating scales will be used to evaluate pain intensity and duration. The pain score (0 min, 20 Max) is derived by adding the numerical rating scores from the pain intensity (0-10, with a score of 0 representing "no pain" and a score of 10 representing "pain as bad as it could be.") and duration scales (0-10, with a score of 0 being "pain none of the time" and a score of 10 being "pain all of the time"). Success for back and leg pain is described as follows:
  Preoperative Score - Postoperative Score >=0
Operative Time | At the time of operation
Blood Loss | At the time of operation
Hospital Days | At the time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Burkus, MD, Principal Investigator — The Hughston Clinic, P.C.; John Dimar, MD, Principal Investigator — Spine Institute
Locations (28):
- United States (28):
  - Barrow Neurosurgical Associates, Phoenix, Arizona
  - Orthopaedic Specialty Institute, Orange, California
  - UCLA Orthopedic Hospital, Santa Monica, California
  - Georgetown University Dept. of Orthopaedic Spine Surgery, Washington D.C., District of Columbia
  - Brevard Orthopaedic Clinic, Inc., Melbourne, Florida
  - Florida Ortho Institute, Tampa, Florida
  - Florida Neurological Consultants, Winter Park, Florida
  - The Hughston Clinic P.C., Columbus, Georgia
  - Barrington Orthopedic Specialists, Hoffman Estates, Illinois
  - Lutheran Spine Center, Park Ridge, Illinois
  - The Spine Institute, Carmel, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Des Moines Orthopaedic Surgeons, West Des Moines, Iowa
  - Spine Institute, Louisville, Kentucky
  - Alvin & Lois Lapidus Cancer Insitute, Baltimore, Maryland
  - Jeffrey S. Fischgrund, Southfield, Michigan
  - Orthopedic Spine Care of Long Island, PC, Melville, New York
  - Beth Israel Medical Center, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Central States Orthopedic Specialists, Tulsa, Oklahoma
  - Medford Neurological & Spine Clinic, Medford, Oregon
  - The Reading Neck & Spine Center, Wyomissing, Pennsylvania
  - East Tennessee Brain & Spine, Johnson City, Tennessee
  - Fort Worth Brain & Spine, Fort Worth, Texas
  - Brain and Spine Center of Texas, Plano, Texas
  - Azalea Orthopedic & Sports Medicine Clinic, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - UVA Dept. of Neurosurgery, Charlottesville, Virginia